CLINICAL TRIAL: NCT03962530
Title: Sarcopenia of Spine: a Prospective Cohort Study
Brief Title: Spinal Sarcopenia Cohort Study (SarcoSpine)
Acronym: SarcoSpine
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Sang Yoon Lee, Clinical associate professor, SMG-SNU Boramae Medical Center
Other Study IDs: 20-2019-19
Record Dates: First submitted 2019-05-21; First posted 2019-05-24 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Sarcopenia; Spinal Disease
MeSH Terms: conditions — Sarcopenia; Spinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sarcopenia on lumbar paraspinal muscles is receiving renewed attention as a cause of spinal degeneration. However, there are few studies on the precise concept and diagnostic criteria for spinal sarcopenia. Here, we develop the concept of spinal sarcopenia in community-dwelling healthy elderly people. In addition, we aim to observe the natural aging course of paraspinal muscle and back muscle strength, and investigate the association between conventional sarcopenic indices and spinal sarcopenia.

This is a prospective observational cohort study with 120 healthy community-dwelling elderly people for 4 years. All subjects will be recruited according to no sarcopenia, possible sarcopenia, sarcopenia, and severe sarcopenia groups. The primary outcomes of this study are isokinetic back muscle strength and lumbar paraspinal muscle quantity and quality using lumbar spine MRI. Conventional sarcopenic indices and spine specific outcomes such as spinal sagittal balance, back performance scale, and Sorenson test will be also assessed. The data will be analysed using the intention-to-treat principle.

DETAILED DESCRIPTION:
This is a prospective observational cohort study with 120 healthy community-dwelling elderly people in a single center (SMG-SNU Boramae Medical Center). Individual follow-up will last 4 years. Elderly people (≥ 65 years old) who are community-dwellers and able to walk with or without assistive devices) will be included. Sarcopenia can be divided by two stages: 1) possible sarcopenia (PS) defined by low handgrip strength and/or low gait speed and 2) sarcopenia (SA) confirmed by low handgrip strength and/or low gait speed and low muscle mass by the consensus report of the Asian working group for sarcopenia. No sarcopenia (NS) group is added to this classification, and the study participants are classified into three groups (NS, PS, and SA) after the screening tests. All outcome variables will be collected at baseline, 2 and 4 years. However, L-S spine MRI for lumbar paraspinal muscle quantity and quality will be performed only at baseline.

Data will be collected using a standardised data entry form and entered into the data management system. The intention-to-treat principle will be used for data analysis. Participant characteristics will be described using means and standard deviations for continuous data and frequencies and percentages for categorical data. The three groups will be compared using an analysis of variance (ANOVA) or the non-parametric equivalence Kruskal-Wallis test if required. To compare paired data (intra-group) between two different points, we will use repeated-measures ANOVA and Friedman tests for continuous and non-parametric data, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Elderly people aged 65 and over;
2. Community dweller;
3. Ambulator with or without an assistive device.

Exclusion Criteria:

1. low back pain with moderate severity (numeric rating scale 5 and over);
2. history of any types of lumbar spine surgery;
3. history of hip fracture surgery and arthroplasty of hip or knee;
4. contraindications for MRI (such as cardiac pacemaker, implanted metallic objects, and claustrophobia);
5. disorders in central nervous system (such as stroke, parkinsonism, spinal cord injury);
6. cognitive dysfunction (Mini Mental State Examination score < 24);
7. communication disorder (such as severe hearing loss);
8. severe cardiopulmonary disease (such as heart failure with New York Heart Association Class III or IV);
9. uncontrolled chronic disease (such as hypertension with systolic blood pressure >165 and diastolic blood pressure >95);
10. musculoskeletal condition affecting physical function (such as amputation of limb);
11. long term use of corticosteroids due to inflammatory disease;
12. malignancy requiring treatment within 5 years; and
13. other medical conditions which needs active treatment; patients who refuse to participate in a study will also be excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Healthy elderly population who are community ambulator.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Change of isokinetic back muscle strength | Baseline, 24 months, and 48 months
  Isokinetic back extensor strength using Biodex
Lumbar paraspinal muscle quantity and quality | Baseline
  Lumbar paraspinal muscle examination using L-S spine MRI

SECONDARY OUTCOMES:
Change of appendicular limb mass | Baseline, 24 months, and 48 months
  Appendicular limb mass measure using wholebody DEXA and BIA
Change of short physical performance battery | Baseline, 24 months, and 48 months
  Physical performance measure by walking speed, balance test, and chair standing
Laboratory test with biomarker | Baseline, 24 months, and 48 months
  Serum IL-6 level
Change of spinal sagittal balance | Baseline, 24 months, and 48 months
  Spinopelvic parameters using simple whole spine X-ray
Change of back performance scale | Baseline, 24 months, and 48 months
  Sock Test, the Pick-up Test, the Roll-up Test, the Fingertip-to-Floor Test, and the Lift Test.

REFERENCES:
- [Derived] Kim JC, Lee SU, Jung SH, Lim JY, Kim DH, Lee SY. Natural aging course of paraspinal muscle and back extensor strength in community-dwelling older adults (sarcopenia of spine, SarcoSpine): a prospective cohort study protocol. BMJ Open. 2019 Sep 5;9(9):e032443. doi: 10.1136/bmjopen-2019-032443. PMID 31492798